CLINICAL TRIAL: NCT07379580
Title: Safety, Reactogenicity, and Immunogenicity of an Mpox mRNA Vaccine Candidate, BNT166a, in Healthy Participants Aged 18 Years and Older in African Countries: A Randomized, Double-blind, Placebo-controlled Phase II Trial
Brief Title: A Randomized Clinical Trial Investigating the Safety, Reactogenicity, and Immunogenicity After Immunization With an mRNA-based Mpox Vaccine Candidate in Africa
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: Coalition for Epidemic Preparedness Innovations (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BNT166-02
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Mpox (Monkeypox); Smallpox; Orthopoxvirus Infection
Keywords: Monkeypox virus (MPXV); Active immunization; Ribonucleic acid (RNA) vaccine
MeSH Terms: conditions — Mpox, Monkeypox; Smallpox; Poxviridae Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1 - BNT166a Dose Level (DL) 1 (Orthopoxvirus-naïve participants, aged 18-45 years) (Experimental): Two doses of investigational medicinal product (IMP).
  Interventions: Biological: BNT166a
- Cohort 1 - BNT166a DL 2 (Orthopoxvirus-naïve participants, aged 18-45 years) (Experimental): Two doses of IMP.
  Interventions: Biological: BNT166a
- Cohort 1 - Placebo (Orthopoxvirus-naïve participants, aged 18-45 years) (Placebo Comparator): 0.9% sodium chloride solution. Two doses of IMP.
  Interventions: Other: Placebo
- Cohort 2 - BNT166a DL 1 (Orthopoxvirus-experienced participants, aged 18-64 years) (Experimental): Two doses of IMP.
  Interventions: Biological: BNT166a
- Cohort 2 - BNT166a DL 2 (Orthopoxvirus-experienced participants, aged 18-64 years) (Experimental): Two doses of IMP.
  Interventions: Biological: BNT166a
- Cohort 2 - Placebo (Orthopoxvirus-experienced participants, aged 18-64 years) (Placebo Comparator): 0.9% sodium chloride solution. Two doses of IMP.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: BNT166a — Intramuscular injection. Injections should be given in the deltoid muscle, using the same non-dominant arm for all IMP doses.
  Arms: Cohort 1 - BNT166a DL 2 (Orthopoxvirus-naïve participants, aged 18-45 years); Cohort 1 - BNT166a Dose Level (DL) 1 (Orthopoxvirus-naïve participants, aged 18-45 years); Cohort 2 - BNT166a DL 1 (Orthopoxvirus-experienced participants, aged 18-64 years); Cohort 2 - BNT166a DL 2 (Orthopoxvirus-experienced participants, aged 18-64 years)
Other: Placebo — Intramuscular injection. Injections should be given in the deltoid muscle, using the same non-dominant arm for all IMP doses.
  Arms: Cohort 1 - Placebo (Orthopoxvirus-naïve participants, aged 18-45 years); Cohort 2 - Placebo (Orthopoxvirus-experienced participants, aged 18-64 years)

SUMMARY:
This is a randomized, double-blind, placebo-controlled study which aims to assess the safety, reactogenicity, and immunogenicity after one and two doses of BNT166a or placebo in healthy participants.

DETAILED DESCRIPTION:
This study will include the following cohorts:

* Cohort 1: healthy adults aged 18 to 45 years inclusive who are Orthopoxvirus-naïve.
* Cohort 2: healthy adults aged 18 to 64 years inclusive who are Orthopoxvirus-experienced.

All participants will receive two doses of BNT166a or placebo at least 28 days apart.

The planned study duration per participant is ~14 months.

ELIGIBILITY:
Key Inclusion Criteria (applicable to all participants unless otherwise specified):

* Are male or female individuals ≥18 years of age at the time of giving informed consent:

  * Cohort 1: ≥18 to ≤45 years of age
  * Cohort 2: ≥18 to ≤64 years of age
* Cohort 1: Participants must be Orthopoxvirus-naïve (have no history of smallpox or mpox vaccination or mpox infection).
* Cohort 2: Participants must be Orthopoxvirus-experienced (have evidence of mpox or smallpox vaccination or mpox infection at least 2 years prior to consent).

Key Exclusion Criteria (applicable to all participants unless otherwise specified):

* Have had recent exposure to mpox (defined as close contact with a probable or confirmed case of mpox within the past 28 days, or have evidence of mpox infection or mpox vaccination within 2 years prior to consent).
* Have a contraindication, warning and/or precaution to vaccination with a messenger ribonucleic acid (mRNA) Coronavirus disease 2019 (COVID-19) vaccine as specified in the Summary of Product Characteristics for BNT162b2 (COMIRNATY United States Prescribing Information/European Union Summary of Product Characteristics) and BNT166 Investigator Brochure.
* Have a history of allergies, hypersensitivities, or intolerance to the study treatments including any excipients thereof.
* Have a current or history of cardiovascular diseases, e.g., myocarditis, pericarditis, myocardial infarction, congestive heart failure, cardiomyopathy, or clinically significant arrhythmias.
* Have any known bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
* Have a body mass index ≤18.5 kg/m^2 or ≥35 kg/m^2.

NOTE: Other protocol defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 310 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Number (and percentage) of participants with at least one solicited local reaction (pain, erythema/redness, induration/swelling) | For up to 7 days following each dose
  At each dose level of BNT166a in Orthopoxvirus-naïve (Cohort 1) and Orthopoxvirus-experienced (Cohort 2) adults.
Number (and percentage) of participants with at least one solicited systemic reaction (fever, headache, fatigue/tiredness, muscle pain/myalgia, joint pain/arthralgia, chills, diarrhea, vomiting) | For up to 7 days following each dose
  At each dose level of BNT166a in Orthopoxvirus-naïve (Cohort 1) and Orthopoxvirus-experienced (Cohort 2) adults.
Number (and percentage) of participants with at least one use of antipyretics/analgesics | For up to 7 days following each dose
  At each dose level of BNT166a in Orthopoxvirus-naïve (Cohort 1) and Orthopoxvirus-experienced (Cohort 2) adults.
Number (and percentage) of participants with at least one unsolicited adverse event (AE) (post-Dose 1) | From Dose 1 to 28 days post-Dose 1
  At each dose level of BNT166a in Orthopoxvirus-naïve (Cohort 1) and Orthopoxvirus-experienced (Cohort 2) adults.
Number (and percentage) of participants with at least one unsolicited AE (post-Dose 2) | From Dose 2 to 28 days post-Dose 2
  At each dose level of BNT166a in Orthopoxvirus-naïve (Cohort 1) and Orthopoxvirus-experienced (Cohort 2) adults.
Number (and percentage) of participants with at least one serious adverse event | From Dose 1 until the end of study, i.e., up to ~14 months
  At each dose level of BNT166a in Orthopoxvirus-naïve (Cohort 1) and Orthopoxvirus-experienced (Cohort 2) adults.
Number (and percentage) of participants with at least one AE of special interest | From Dose 1 until the end of study, i.e., up to ~14 months
  At each dose level of BNT166a in Orthopoxvirus-naïve (Cohort 1) and Orthopoxvirus-experienced (Cohort 2) adults.
Number (and percentage) of participants with at least one medically attended AE | From Dose 1 until the end of study, i.e., up to ~14 months
  At each dose level of BNT166a in Orthopoxvirus-naïve (Cohort 1) and Orthopoxvirus-experienced (Cohort 2) adults.
Number (and percentage) of participants with at least one AE leading to a participant's withdrawal from the study | From Dose 1 until the end of study, i.e., up to ~14 months
  At each dose level of BNT166a in Orthopoxvirus-naïve (Cohort 1) and Orthopoxvirus-experienced (Cohort 2) adults.

SECONDARY OUTCOMES:
Geometric mean titers (GMT) of BNT166a antigen-specific (A35, B6, H3, and M1) binding antibody titers | At baseline, 1 month post-Dose 1, and 1 month post- Dose 2
  At each dose level of BNT166a in Orthopoxvirus-naïve (Cohort 1) and Orthopoxvirus-experienced (Cohort 2) adults, at the defined timepoints.
Geometric mean fold rise (GMFR) of BNT166a antigen-specific (A35, B6, H3, and M1) binding antibody titers | At 1 month post-Dose 1 and 1 month post-Dose 2
  At each dose level of BNT166a in Orthopoxvirus-naïve (Cohort 1) and Orthopoxvirus-experienced (Cohort 2) adults.
  Ratio post-baseline/baseline at the defined timepoints.
GMT of MPXV-specific neutralizing antibody titers | At baseline, 1 month post-Dose 1, and 1 month post-Dose 2
  At each dose level of BNT166a in Orthopoxvirus-naïve (Cohort 1) and Orthopoxvirus-experienced (Cohort 2) adults, at the defined timepoints.
GMFR of MPXV-specific neutralizing antibody titers | At 1 month post-Dose 1 and 1 month post-Dose 2
  At each dose level of BNT166a in Orthopoxvirus-naïve (Cohort 1) and Orthopoxvirus-experienced (Cohort 2) adults.
  Ratio post-baseline/baseline at the defined timepoints.
GMT of vaccinia virus (VACV)-specific neutralizing antibody titers | At baseline, 1 month post-Dose 1, and 1 month post-Dose 2
  At each dose level of BNT166a in Orthopoxvirus-naïve (Cohort 1) and Orthopoxvirus-experienced (Cohort 2) adults, at the defined timepoints.
GMFR of VACV-specific neutralizing antibody titers | At 1 month post-Dose 1 and 1 month post-Dose 2
  At each dose level of BNT166a in Orthopoxvirus-naïve (Cohort 1) and Orthopoxvirus-experienced (Cohort 2) adults.
  Ratio post-baseline/baseline at the defined timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (6):
- Democratic Republic of the Congo (2):
  - University of Kinshasa UNIKIN, Kinshasa
  - Institute National de Recherche Biomedicale, Kinshasa
- South Africa (4):
  - TASK Applied Science, Cape Town
  - TREAD Research Pty Ltd, Cape Town
  - Desmond Tutu Health Foundation Masiphumelele Clinic, Cape Town
  - Perinatal HIV Research Unit, Johannesburg

IPD SHARING:
Plan to Share IPD: No